CLINICAL TRIAL: NCT05813379
Title: Application of Mesenchymal Stem Cells Derived Exosomes in Skin Rejuvenation
Brief Title: Mesenchymal Stem Cells Derived Exosomes in Skin Rejuvenation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Leila Dehghani, Principal Investigator, Isfahan University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Islamic Azad University
Record Dates: First submitted 2022-12-26; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Anti Aging
Keywords: Anti aging; Rejuvenation; Repair; Regeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- exosome injection (Experimental): The Exosome will be injected into each standardized injection point in a superficial manner. The injections points are along the inferior border of cheek and mid-cheek and temple, where will be followed by 10-15 minutes of icing
  Interventions: Combination Product: exosime injection

INTERVENTIONS:
Combination Product: exosime injection — Treatment- exosome injection

SUMMARY:
Aging is a natural and complex process. The effect of environmental factors, genetics on the body eventually leads to damage in different ways. Exosomes are present in almost all body fluids, such as synovial fluid and blood. Exosomes and microvesicles are very efficient mediators of cell-to-cell communication by transferring their specific cargo to recipient cells; for example, exosomes are involved in the delivery of genetic materials, causing epigenetic modifications in the target cells .The applications of MSC-derived exosomes have more effect in cutaneous regeneration by collagen stimulation.The basic biology of exosomes indicates that MSC-exosomes may contain MSC-specific components to exert specific effects on recipient cells, which are somewhat equivalent to the regenerative effects of MSCs. This study aims to slow down the aging process of the skin by using exosome.

DETAILED DESCRIPTION:
Skin aging is a complex biological process that can be classified into extrinsic or intrinsic aging. Intrinsic aging is an intrinsic degradation process that is caused by a decrease in the proliferation capacity leading to cell senescence. Angiogenesis is essential in various physiological processes, including wound healing and skin tissue regeneration. Literature reviews show that exosomes derived from human umbilical cord blood mesenchymal stem cells can cause Collagen stimulation and reduction of oxidative stress, WNT/βcatenin pathway signaling in the initial stages of causes the regeneration of skin damage . This study aims to slow down the aging process of the skin by using exosome.

ELIGIBILITY:
Inclusion Criteria:

* females
* Ages 35-65
* Patients of all racial and ethnic origins
* Patients of all undergoing facial rejuvenation

Exclusion Criteria:

* Female patients in pregnancy or menstrual period
* Patients undergoing facial rejuvenation using other methods including Botox injections, chemical peels, face lifts and others
* Patients using blood thinners, aspirin and hormone, that cannot be stopped
* Patients suffering with severe organic disease, such as coronary heart disease, hypertension, diabetes, lung dysfunction and so on
* Patients suffering with mental disease, and acute or chronic infectious diseases

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-07-29 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of re-epithelialization | 1 month
  In order to evaluate the treatment effect, to evaluate wrinkles and collagen before the treatment, take a photo/CT of the face
Proportion of re-epithelialization | 3 months
  In order to evaluate the treatment effect, to evaluate wrinkles and collagen before the treatment, take a photo/CT of the face

CONTACTS AND LOCATIONS:
Overall Officials: Leila Dehghani, Principal Investigator — university of medical sciences
Locations (1):
- Isfahan University of Medical Sciences, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Undecided